CLINICAL TRIAL: NCT00188838
Title: Psychoeducation Versus Cognitive-Behavioral Therapy in Bipolar Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Stanley Medical Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 02-0378-E
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2005-09-16 (Estimated); Status verified 2005-07

CONDITIONS: Bipolar Disorder
Keywords: Bipolar Disorder; Psychosocial Factors; Mania; Depression; Social Adjustment; Coping Skills
MeSH Terms: conditions — Bipolar Disorder; Mania; Depression; Social Adjustment | interventions — Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Psychoeduction
Behavioral: Cognitive-Behavioral Therapy

SUMMARY:
To examine the impact of cognitive-behavioural therapy on both the episodic and functional outcome of bipolar disorder, in combination with pharmacotherapy.

Primary Hypothesis is twofold:

1. Cognitive Behavioural Therapy will reduce the total symptom burden, as measured both by percentage of time spent ill (both syndromic and subsyndromal) and number of episodes, as compared to psychoeducation
2. Cognitive behavioural therapy will reduce social and occupational disability to a greater extent than psychoeducation.

DETAILED DESCRIPTION:
Objective:

To compare the impact of cognitive -behavioral therapy to that of properly structured psycho education on the 'illness burden' and functional outcome of bipolar disorder, in combination with pharmacotherapy.

Interventions:

Subjects will be randomized to either a "control" treatment group cosisting of 6 sessions of group psycho-education (topics include illness recognition, treatment approaches, and monitoring and coping strategies; based on manual by Bauer & McBride, 2002: Life Goals Phase I) or they will be randomized to the "experimental" treatment group: 20 sessions of individual Cognitive Behavioural Therapy for Bipolar Disorder (topics include limited psychoeducation, activity scheduling/behavioural interventions, cognitive techniques, including thought monitoring and challenges to dysfunctional assumptions and other coping techniques; based on manual by Lam et al., 1999: Cognitive Therapy for Bipolar Disorder)

ELIGIBILITY:
Inclusion Criteria:

1. Bipolar I or II
2. Currently either in remission or subsyndromally ill (Hamilton Depression Scale-17<14; Clinician Administered Rating Scale for Mania<12).
3. Age eighteen to sixty.
4. Significant symptoms and/or episodes on at least two occasions in the past three years.
5. Grade six education, able to understand English, and Folstein Minimental Score Exam > 26 to ensure cognitive ability to participate.
6. On mood-stabilizing medication.

Exclusion Criteria:

1. Substance dependence meeting Diagnostic and Statistical Manual of Mental Disorders-IV criteria within the last three months.
2. Acutely highly suicidal or homicidal.
3. Serious other medical condition that would render pharmacotherapy or psychotherapy very difficult such as cancer, severe diabetes, etc.
4. Severe antisocial or borderline personality disorder (personality disorder per se is not exclusionary). Subjects may have other axis I disorders, but bipolar disorder must be the principal disorder requiring treatment.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 210
Dates: Start 2002-07; Study Completion 2006-08

PRIMARY OUTCOMES:
Longitudinal Interval Follow-up Evaluation (LIFE; Keller et al, 1987).
Modified Social Adjustment Scale (SAS II-B; Bauer, 2001)
***Note: all primary outcomes obtained prospectively every 3 months for 18 months

SECONDARY OUTCOMES:
Clinician Administered Rating Scale for Mania
Hamilton Depression Rating Scale
Quality of Life, Enjoyment, and Satisfaction Questionnaire
Dysfunctional Attitudes Scale
Patient Satisfaction Index
Activity and Utilisation Questionnaire
Medication Compliance scale
Intensity of Somatotherapy Index
Coping Inventory for Prodromes of Mania
Khavari Alcohol Test.
*****Note: all secondary outcomes measured prospectively over 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Sagar V Parikh, M.D., Principal Investigator — University Health Network, Toronto
Locations (6):
- Canada (6):
  - University of British Columbia, Department of Psychiatry, Vancouver, British Columbia
  - St. Joseph's Healthcare, CMHS, Hamilton, Ontario
  - Centre for Addiction and Mental Health, Toronto, Ontario
  - University Health Network, Toronto, Ontario
  - McGill University Health Centre, Montreal, Quebec
  - Douglas Hospital-McGill University, Verdun, Quebec

REFERENCES:
- [Derived] Parikh SV, Hawke LD, Velyvis V, Zaretsky A, Beaulieu S, Patelis-Siotis I, MacQueen G, Young LT, Yatham LN, Cervantes P. Combined treatment: impact of optimal psychotherapy and medication in bipolar disorder. Bipolar Disord. 2015 Feb;17(1):86-96. doi: 10.1111/bdi.12233. Epub 2014 Jul 21. PMID 25046246
- [Derived] Parikh SV, Hawke LD, Zaretsky A, Beaulieu S, Patelis-Siotis I, Macqueen G, Young LT, Yatham L, Velyvis V, Belanger C, Poirier N, Enright J, Cervantes P. Psychosocial interventions for bipolar disorder and coping style modification: similar clinical outcomes, similar mechanisms? Can J Psychiatry. 2013 Aug;58(8):482-6. doi: 10.1177/070674371305800807. PMID 23972110
- [Derived] Parikh SV, Zaretsky A, Beaulieu S, Yatham LN, Young LT, Patelis-Siotis I, Macqueen GM, Levitt A, Arenovich T, Cervantes P, Velyvis V, Kennedy SH, Streiner DL. A randomized controlled trial of psychoeducation or cognitive-behavioral therapy in bipolar disorder: a Canadian Network for Mood and Anxiety treatments (CANMAT) study [CME]. J Clin Psychiatry. 2012 Jun;73(6):803-10. doi: 10.4088/JCP.11m07343. PMID 22795205